CLINICAL TRIAL: NCT05575284
Title: Pain Intensity After RObotic Assisted Urological Surgery: the PAIROU Study
Brief Title: Pain Intensity After RObotic Assisted Urological Surgery
Acronym: PAIROU
Status: Completed | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: PAIROU 2022-04
Record Dates: First submitted 2022-09-29; First posted 2022-10-12 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Robot-assisted Urological Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Robot-assisted urological surgery: Patients with programmed robot-assisted urological surgery
  Interventions: Procedure: Robot-assisted urological surgery

INTERVENTIONS:
Procedure: Robot-assisted urological surgery — Patient with programmed robot-assisted urological surgery

SUMMARY:
Postoperative pain remains a widespread but still underestimated problem. Studies have shown that despite improvements in pain management, many patients still suffer from moderate to severe postoperative pain. Severe pain is associated with decreased patient satisfaction, delayed postoperative ambulation, prolonged length of stay, risk of developing chronic postoperative pain, and increased morbidity and mortality. Therefore, it is of great importance that surgical procedures that result in severe pain and the optimal analgesic strategies for these procedures can be identified. Most recommendations on postoperative pain management (prevention and treatment) are not procedure-specific. However, risk factors for postoperative pain depend on the patient and the procedure.

In order to develop procedure-specific postoperative pain management guidelines, pain must be assessed in a procedure-specific manner. Additionally, data is sparse on relatively new procedures like robotic surgery. A study, Harel et al. compared pain intensities after ureteral reimplantation with robotic or open surgery in children and reported lower pain scores after robotic surgery. This single study reinforces the clinical findings that robotic surgery is associated with less pain. However, pain assessment after robotic urologic surgery has not been evaluated before.

In order to add to the evaluation of postoperative pain in different surgical groups, we wish to evaluate pain intensities after robot-assisted urological surgery. In this cohort study, we seek to provide an estimate of the pain intensities that can be expected after most types of robot-assisted urological surgery in relation to analgesic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Programmed robot-assisted urological surgery
* Patient who did not declare any opposition to participating in the study

Exclusion Criteria:

* Urgent surgery
* Impossibility of communicating in French
* Cognitive deficit
* Adults legally protected or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with planned robot-assisted urological surgery.
Sampling Method: Non-Probability Sample
Enrollment: 968 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Pain level on D1 of surgery | Day 1 after surgery
  Measurement of pain intensity on D1 of surgery, assessed with a simple numerical scale (ENS). Scores range from 0-10 points, with higher scores indicating greater pain intensity.

SECONDARY OUTCOMES:
Pain intensity (NRS) at rest and during exercise | Second day after surgery
  Pain intensity on the second day after surgery (NRS) at rest and during exercise. Pain intensity assessed with a simple numerical scale (ENS). Scores range from 0-10 points, with higher scores indicating greater pain intensity.
Highest pain score at rest and during exercise | In the first 48 hours
  Highest pain score in the first 48 hours at rest and during exercise. Pain intensity assessed with a simple numerical scale (ENS). Scores range from 0-10 points, with higher scores indicating greater pain intensity.
Presence of side effect: Nausea and vomiting | In the first 48 hours
  Patient presenting or not nausea and vomiting in the first 48 hours
Time of the first ambulation | Time of the first ambulation during hospitalization
  Time from robotic assisted urological surgery to the first ambulation
Date and time of resumption of transit | Date and time of resumption of transit
  number of days between robotic assisted urological surgery and resumption of transit
Consumption of morphine | During the 48 hours after surgery
  Consumption of morphine (or equivalent (see morphine equivalent table)) in mg 48 hours after surgery
Duration of surgery | Duration of surgery
  Duration of surgery: time between the begining of the robotic assisted urological surgery and the end of surgery.
Operator experience for the robotic assisted urological surgery | Operator experience is the number of years from the first robotic assisted urological surgery performed by the operator until the surgery of the patient included in this study.
  Operator experience for the robotic assisted urological surgery, classified in 3 ranges: less than 5 years; between 5 and 10 years; more than 10 years
Complications | Period is defined from the day of robotic assisted urological surgery until the end of hospitalisation
  Complications according to the Dindo and Clavien classification
Length of stay | From the first day of hospitalization to the last day of hospitalization
  Length of stay at hospital (number of days)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BELOEIL, MD, Study Chair — Teaching Hospital of Rennes, France
Locations (46):
- CHU St Pierre - Bruxelles, Brussels, Belgium
- France (43):
  - Clinique Victor PAUCHET, Amiens
  - Clinique de l'Anjou, Angers
  - Hôpital Privé Arras les Bonnettes, Arras
  - Polyclinique Sainte Marguerite - Institut d'Urologie- Auxerre, Auxerre
  - Hôpital Privé de la Châtaigneraie - Beaumont, Beaumont
  - Clinique Saint Vincent, Besançon
  - CH de Bourg en Bresse, Bourg-en-Bresse
  - Centre Hospitalier Dubois - Brive la Gaillarde, Brive-la-Gaillarde
  - CH de Dax, Dax
  - CHU Grenoble Alpes, La Tronche
  - Hopital Bicêtre - APHP, Le Kremlin-Bicêtre
  - Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille
  - Hôpital Huriez - CHU de Lille, Lille
  - Hôpital Edouard Herriot (HCL - Lyon), Lyon
  - CH Saint Joseph Saint Luc, Lyon
  - Hôpital Privé Jean Mermoz - Lyon, Lyon
  - CHU Conception - Marseille, Marseille
  - Hôpital Nord de Marseille, Marseille
  - CH de Mont-de-Marsan, Mont-de-Marsan
  - CHU de Nantes, Nantes
  - GH Privé Ambroise Paré - Hartmann, Neuilly-sur-Seine
  - CHU de Nimes-Hôpital Carémeau, Nîmes
  - CHR Orléans, Orléans
  - Hôpital Saint-Louis - APHP, Paris
  - AP-HP - Groupe Hospitalier Pitié-Salpêtrière - APHP, Paris
  - Hôpital Bichat - APHP, Paris
  - Hôpital Tenon - APHP, Paris
  - CH Perpignan, Perpignan
  - CHU Guadeloupe, Pointe à Pitre
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU Réunion (site Nord), Saint-Denis
  - CH de Saintonge, Saintes
  - CH de Seclin, Seclin
  - CH de Sens, Sens
  - Centre Clinical - Soyaux, Soyaux
  - Clinique Rhéna - Strasbourg, Strasbourg
  - Clinique Sainte Anne, Strasbourg
  - Hôpital Foch, Suresnes
  - Centre Hospitalier Intercommunal Toulon-La Seyne sur mer, Toulon
  - CHU Toulouse - Hôpital Rangueil, Toulouse
  - CH de Valenciennes, Valenciennes
  - CHRU de Nancy, Vandœuvre-lès-Nancy
- Spain (2):
  - Hospital Universitario La Zarzuela, Madrid
  - Hospital Clínico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Aubrun F, Nouette-Gaulain K, Fletcher D, Belbachir A, Beloeil H, Carles M, Cuvillon P, Dadure C, Lebuffe G, Marret E, Martinez V, Olivier M, Sabourdin N, Zetlaoui P. Revision of expert panel's guidelines on postoperative pain management. Anaesth Crit Care Pain Med. 2019 Aug;38(4):405-411. doi: 10.1016/j.accpm.2019.02.011. Epub 2019 Feb 26. PMID 30822542
- [Background] Panzenbeck P, von Keudell A, Joshi GP, Xu CX, Vlassakov K, Schreiber KL, Rathmell JP, Lirk P. Procedure-specific acute pain trajectory after elective total hip arthroplasty: systematic review and data synthesis. Br J Anaesth. 2021 Jul;127(1):110-132. doi: 10.1016/j.bja.2021.02.036. PMID 34147158
- [Background] Harel M, Herbst KW, Silvis R, Makari JH, Ferrer FA, Kim C. Objective pain assessment after ureteral reimplantation: comparison of open versus robotic approach. J Pediatr Urol. 2015 Apr;11(2):82.e1-8. doi: 10.1016/j.jpurol.2014.12.007. Epub 2015 Feb 26. PMID 25864615
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Derived] Rouxel P, Rayon E, Bellocq AS, le Guen M, Fessler J, Cirenei C, Blondonnet R, Parfait E, Patrubani AG, Ramorasata A, Gouel A, Brogly N, Devoldere G, Dupont M, Gaultier E, Dupuis M, Bouzat P, Cattenoz M, Prieur S, Cuvillon P, Gricourt Y, Pastene B, Huette P, Garot M, Ramarosaona A, Massin R, Grailles G, Rolle A, Daouda IM, Boinette R, Birckener J, Habrial P, Samaha T, Lemoine A, Damon A, Rodriguez M, Braun T, Fritsch M, Tawil S, Guerin V, Lagrave-Blampied L, Ravry C, Poette M, Tao-Mauny S, Mfam WS, Fontaine M, Boutouria M, Deffar N, Sigwalt F, Thiltges L, Ionescu M, Diaz-Pache MVA, Perez RN, Caragliano G, Profumo L, Peyronnet B, Renault A, Joosten A, Beloeil H; PAIROU group and French Society of Anesthesiologists (SFAR) Research Network. Pain intensity after robotic-assisted urological surgery: the PAIROU study an international prospective cohort study. Anaesth Crit Care Pain Med. 2025 Aug;44(4):101546. doi: 10.1016/j.accpm.2025.101546. Epub 2025 May 21. PMID 40409579